CLINICAL TRIAL: NCT03662256
Title: Addressing Early Childhood Hearing Loss in Rural Alaska: A Community Randomized Trial
Brief Title: Reducing Childhood Hearing Loss in Rural Alaska Through a Preschool Screening and Referral Process Using Mobile Health and Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norton Sound Health Corporation (Other)
Collaborators: Duke University (Other); Johns Hopkins University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AD-1602-34571-S1
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Hearing Loss
Keywords: hearing loss; deafness; hearing disorders; ear diseases; otorhinolaryngologic diseases; child, preschool
MeSH Terms: conditions — Hearing Loss; Deafness; Hearing Disorders; Ear Diseases; Otorhinolaryngologic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The randomization assignments will be kept confidential within the study team until hearing screening day, when masking the referral process assignment to participants will no longer be possible. All outcome assessors, including audiologists and ear, nose, and throat (ENT) surgeons reading telemedicine consults within the Alaska Native healthcare system and study team members performing medical record abstraction, will be masked to intervention allocation throughout the trial. Study team members who read telemedicine consults as a part of their clinical responsibilities will abstain from reading any study-related consults. The results of the preschool screen, mHealth screen, and audiometric assessments will also be masked, such that study team members performing the mHealth screen or audiometric assessment will be masked to the other results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current Primary Care Referral Process (Active Comparator): In communities randomized to the current primary care process, families will be notified if their children refer hearing screening in exactly the same method each preschool had been using previously. This process involves a letter home to the parents, either sent with the child or by mail, requesting that the parent/caregiver bring the child to village health clinic for an evaluation. Per current practice, most preschools also give the list of referred children to the Norton Sound Audiology Department, whose staff then reaches out to families to schedule appointments during the next available audiology clinic.
  Interventions: Other: Current Primary Care Referral Process
- Expedited Telemedicine Referral (Experimental): In communities randomized to the expedited telemedicine intervention, parents of children who screen positive will receive a phone call from the school or the clinic on the day of screening notifying them of the day and time of their child's telemedicine consultation appointment. Appointments will be made with community health aides (CHAs) who have dedicated time blocked off to perform telemedicine consults. Participating children who refer screening will be transported to clinic for their appointment with adult chaperones. Parent participation will be required unless parents direct otherwise. Nonparticipating children in communities assigned to the expedited telemedicine intervention arm will receive standard referral following the current school primary care referral process.
  Interventions: Other: Telemedicine Referral Process

INTERVENTIONS:
Other: Current Primary Care Referral Process — Children who refer hearing screening will receive the same referral method each preschool had been using previously. This process involves a letter home to the parents, either sent with the child or by mail, requesting that the parent/caregiver bring the child to village health clinic for an evaluation.
  Arms: Current Primary Care Referral Process
Other: Telemedicine Referral Process — In communities randomized to the expedited telemedicine intervention, parents of children who refer hearing screening will receive a phone call from the school or the clinic on the day of screening notifying them of the day and time of their child's telemedicine consultation appointment. Appointments will be made with community health aides (CHAs) who have dedicated time blocked off to perform telemedicine consults. Participating children who refer screening will be transported to clinic for their appointment with adult chaperones. Parent participation will be required unless parents direct otherwise. Nonparticipating children in communities assigned to the expedited telemedicine intervention arm will receive standard referral following the current school primary care referral process.
  Arms: Expedited Telemedicine Referral

SUMMARY:
The population in rural Alaska, which is predominately Alaska Native, experiences a disproportionately high burden of hearing loss compared to the general US population. The impact of untreated hearing loss in early childhood is tremendous and has grave implications for school achievement. Preschool children with hearing loss experience speech and language delays and are less likely to be ready for kindergarten than their normal-hearing peers. Early identification and treatment can reverse these ill effects. Importantly, the majority of hearing loss in this age group in rural Alaska is infection-mediated, arising from acute and chronic otitis media that is treatable.

In response, preschool hearing screening is federally mandated at all Head Start centers across the country. In accordance with this mandate, hearing screening is already performed by the three organizations that offer early childhood education in the Norton Sound region: Kawerak Inc, RurAL CAP, and Bering Strait School District.

While the concept of screening in this age group is well established nationally, what is less well understood is the optimal screening protocol for preschool children. There is little evidence evaluating sensitivity and specificity of different screening protocols in this age group. Further, loss to follow up in the referral stage is a problem in preschool hearing screening just as it is in school hearing screening.

Alaska has already developed innovative strategies to address hearing loss. A network of village health clinics staffed by community health aides provide local care, and telemedicine has been adopted in over 250 village clinics statewide. Despite being widely available, telemedicine has not yet been used to speed up the referral process for preventive services such as hearing screening.

Norton Sound Health Corporation has partnered with Duke and Johns Hopkins Universities to evaluate hearing screening and referral processes in early childhood education in the Norton Sound region of northwest Alaska. Preschool children will receive screening from the preschool and a new mHealth screening protocol. These will be compared against a benchmark audiometric assessment to determine sensitivity and specificity. Communities will then be randomized to continue the current primary care referral process or to adopt telemedicine referral. The primary outcome will be time to ICD-10 ear/hearing diagnosis. Secondary outcomes will include sensitivity and specificity of screening protocols and prevalence of hearing loss. The goal of this study is to evaluate the optimal screening and referral strategy for preschool children in rural Alaska.

ELIGIBILITY:
Inclusion Criteria:

* Early childhood education student of the Bering Strait School District (BSSD), Kawerak Inc, or RurAL CAP in the Norton Sound region of Northwest Alaska
* All preschool-aged children, enrolled in one of the three organizations that provide early childhood education in the region, are eligible to participate
* Parental signed consent to undergo routine hearing screening in the preschool setting
* Child assent from children enrolled in the study

Exclusion Criteria:

* Not an early education student of the Bering Strait School District, Kawerak Inc, or RurAL CAP.
* Parental consent for routine hearing screening not obtained
* Child assent not obtained

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Time to diagnosis | From date of screening to date of ICD-10 ear/hearing diagnosis, measured in days, up to 9 months from date of screening
  Comparing time to International Classification of Disease, Tenth Edition (ICD-10) ear/hearing diagnosis from date of screening between intervention and active comparator

SECONDARY OUTCOMES:
Sensitivity and specificity of screening protocols | Cross-sectional comparison of concurrent mHealth screening protocol and current preschool hearing screening to audiometric assessment, measured once in the 2018-2019 academic year, all communities combined
  School and mobile health (mHealth) screening to audiometric assessment, all measured on the same day in Baseline before intervention
Prevalence of hearing loss | Baseline before intervention
  Estimating baseline prevalence of hearing loss in preschool children using audiometric assessments, all communities combined

CONTACTS AND LOCATIONS:
Locations (1):
- Norton Sound Health Corporation, Nome, Alaska, United States

REFERENCES:
- [Derived] Jin FQ, Huang O, Kleindienst Robler S, Morton S, Platt A, Egger JR, Emmett SD, Palmeri ML. A Hybrid Deep Learning Approach to Identify Preventable Childhood Hearing Loss. Ear Hear. 2023 Sep-Oct 01;44(5):1262-1270. doi: 10.1097/AUD.0000000000001380. Epub 2023 Jun 15. PMID 37318215
- [Derived] Emmett SD, Platt A, Gallo JJ, Labrique AB, Wang NY, Inglis-Jenson M, Jenson CD, Hofstetter P, Hicks KL, Ross AA, Egger JR, Robler SK. Prevalence of Childhood Hearing Loss in Rural Alaska. Ear Hear. 2023 Sep-Oct 01;44(5):1240-1250. doi: 10.1097/AUD.0000000000001368. Epub 2023 Jun 8. PMID 37287104
- [Derived] Robler SK, Platt A, Turner EL, Gallo JJ, Labrique A, Hofstetter P, Inglis-Jenson M, Jenson CD, Hicks KL, Wang NY, Emmett SD. Telemedicine Referral to Improve Access to Specialty Care for Preschool Children in Rural Alaska: A Cluster-Randomized Controlled Trial. Ear Hear. 2023 Nov-Dec 01;44(6):1311-1321. doi: 10.1097/AUD.0000000000001372. Epub 2023 May 25. PMID 37226299
- [Derived] Robler SK, Platt A, Jenson CD, Meade Inglis S, Hofstetter P, Ross AA, Wang NY, Labrique A, Gallo JJ, Egger JR, Emmett SD. Changing the Paradigm for School Hearing Screening Globally: Evaluation of Screening Protocols From Two Randomized Trials in Rural Alaska. Ear Hear. 2023 Jul-Aug 01;44(4):877-893. doi: 10.1097/AUD.0000000000001336. Epub 2023 Mar 13. PMID 36907833
- [Derived] Hicks KL, Robler SK, Platt A, Morton SN, Egger JR, Emmett SD. Environmental Factors for Hearing Loss and Middle Ear Disease in Alaska Native Children and Adolescents: A Cross-Sectional Analysis from a Cluster Randomized Trial. Ear Hear. 2023 Jan-Feb 01;44(1):2-9. doi: 10.1097/AUD.0000000000001265. Epub 2022 Aug 23. PMID 35998103